CLINICAL TRIAL: NCT03702621
Title: Liposomal Bupivacaine Versus Standard Bupivacaine Hydrochloride In Colorectal Surgery
Brief Title: Comparing Liposomal Bupivacaine Versus Standard Bupivacaine in Colorectal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Yar Yeap, Director, Acute Pain Service Assistant Professor of Clinical Anesthesiology Indiana University School of Medicine Department of Anesthesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1806187876
Record Dates: First submitted 2018-08-06; First posted 2018-10-11 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Surgery
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: 1. LB group (Liposomal Bupivacaine)
  2. SB group (Standard Bupivacaine)
Who Masked: Participant, Investigator
Masking Description: Both the patients and the research staff doing assessments will be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine (Active Comparator): LB (Liposomal Bupivacaine) group - This group will be receiving 20 mL EXPAREL (266mg) and 40 mL of 0.125% bupivacaine in total, 30ml on each side.
  For the QL block, Shamrock sign consistent of the quadratus lumborum muscle, psoas major muscle, erector spinae muscles and the L4 transverse process will be identified. Under ultrasound guidance with an in-plane technique, the needle will be advanced into the fascial plane between the quadratus lumborum and psoas major muscles. Local anesthetic will be injected into the plane.
  Interventions: Drug: liposomal Bupivacaine
- Standard Bupivacaine (Active Comparator): SB (Standard Bupivacaine) group - This group will be receiving 60 mL of 0.25% bupivacaine in total, 30 mL on each side.
  For the QL block, Shamrock sign consistent of the quadratus lumborum muscle, psoas major muscle, erector spinae muscles and the L4 transverse process will be identified. Under ultrasound guidance with an in-plane technique, the needle will be advanced into the fascial plane between the quadratus lumborum and psoas major muscles. Local anesthetic will be injected into the plane.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: liposomal Bupivacaine — 20 mL liposomal bupivacaine are injected into the liposomal bupivacaine group
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine Hydrochloride — 40 mL of 0.125% bupivacaine hydrochloride are injected into the liposomal bupivacaine group.
  60mL of 0.25% bupivacaine hydrochloride are injected into the standard bupivacaine group
  Arms: Standard Bupivacaine

SUMMARY:
The purpose of this study is to compare the difference between two different pain control methods in patients who will be having a colorectal surgery

DETAILED DESCRIPTION:
Quadratus lumborum (QL) blocks will be done intraoperatively after induction. All procedures will be placed under the supervision of the attending anesthesiologist on the acute pain service.

All patients will receive 1 gm acetaminophen and 600 mg gabapentin preoperatively. Patients above 70yo will receive 300mg gabapentin. Patient will be randomized to one of the two arms.

For the QL block, Shamrock sign consistent of the quadratus lumborum muscle, psoas major muscle, erector spinae muscles and the L4 transverse process will be identified. Under ultrasound guidance with an in-plane technique, the needle will be advanced into the fascial plane between the quadratus lumborum and psoas major muscles. For the liposomal bupivacaine (LB) group, 0.125% bupivacaine 20ml plus Exparel®10ml will then be injected into the fascial plane on each side. For the standard bupivacaine (SB) group. 30ml 0.25% bupivacaine will be injected on each side. Saline will be used for hydro-dissection until the QL block target is confirmed on ultrasound.

As part of the enhanced recovery after surgery (ERAS) protocol, all patients will receive ketamine and lidocaine drip during surgery, which is the investigator's current standard of practice.

All patients will be scheduled on PO acetaminophen and PO gabapentin daily postoperatively per ERAS protocol. PO oxycodone as needed (PRN) will be started once patients tolerate diet. PRN IV dilaudid may be given for severe breakthrough pain.

Opioid usage at 1, 24, 48 and 72 hours after the block will be recorded by a member of the research team. Pain scores at rest and on movement (knee flexion) will be measured by the investigator using Visual Analog Scale (VAS). Nausea will be measured using a categorical scoring system (none=0; mild=1; moderate=2; severe=3). Sedation scores will also be assessed by a member of the study team using a sedation scale (awake and alert=0; quietly awake=1; asleep but easily roused=2; deep sleep=3). All these parameters will be measured at 1, 24, 48 and 72 hours after the QL block and patients will be encouraged to ambulate on postoperative day 1 under supervision. Their ambulation activity will be recorded.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing colorectal surgery at Indiana University Hospital
* American Society of Anesthesiologists (ASA) class 1, 2, 3 or 4
* Age 18 or older, male or female
* Desires Regional anesthesia for postoperative pain control

Exclusion criteria:

* Any contraindication for QL block.
* History of substance abuse in the past 6 months.
* Patients on more than 30mg morphine equivalents of opioids daily.
* Any physical, mental or medical conditions which in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery.
* Known allergy or other contraindications to the study medications (Acetaminophen, Gabapentin, Bupivacaine).
* Postoperative intubation.
* Any BMI greater than 40.0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yar Yeap, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Yeap YL, Wolfe J, Stewart J, McCutchan A, Chawla G, Robb B, Holcomb B, Vickery B. Liposomal bupivacaine addition versus standard bupivacaine alone for colorectal surgery: a randomized controlled trial. Pain Manag. 2022 Jan;12(1):35-43. doi: 10.2217/pmt-2021-0033. Epub 2021 Sep 23. PMID 34551581

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine: LB (Liposomal Bupivacaine) group - This group will be receiving 20ml EXPAREL (266mg) and 40ml of 0.125% bupivacaine in total, 30ml on each side.
  For the QL block, Shamrock sign consistent of the quadratus lumborum muscle, psoas major muscle, erector spinae muscles and the L4 transverse process will be identified. Under ultrasound guidance with an in-plane technique, the needle will be advanced into the fascial plane between the quadratus lumborum and psoas major muscles. Local anesthetic will be injected into the plane.
  liposomal Bupivacaine: 20mL liposomal bupivacaine are injected into the liposomal bupivacaine group
- Standard Bupivacaine: SB (Standard Bupivacaine) group - This group will be receiving 60ml of 0.25% bupivacaine in total, 30ml on each side.
  For the QL block, Shamrock sign consistent of the quadratus lumborum muscle, psoas major muscle, erector spinae muscles and the L4 transverse process will be identified. Under ultrasound guidance with an in-plane technique, the needle will be advanced into the fascial plane between the quadratus lumborum and psoas major muscles. Local anesthetic will be injected into the plane.
  Bupivacaine Hydrochloride: 40ml of 0.125% bupivacaine hydrochloride are injected into the liposomal bupivacaine group.
  60mL of 0.25% bupivacaine hydrochloride are injected into the standard bupivacaine group
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Started | 44 | 46
Completed | 38 | 40
Not Completed | 6 | 6
Not completed — Physician Decision | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Liposomal Bupivacaine: LB (Liposomal Bupivacaine) group - This group will be receiving 20 mL EXPAREL (266mg) and 40 mL of 0.125% bupivacaine in total, 30 mL on each side.
  For the quadratus lumborum (QL) block, Shamrock sign consistent of the quadratus lumborum muscle, psoas major muscle, erector spinae muscles and the L4 transverse process will be identified. Under ultrasound guidance with an in-plane technique, the needle will be advanced into the fascial plane between the quadratus lumborum and psoas major muscles. Local anesthetic will be injected into the plane.
  liposomal Bupivacaine: 20 mL liposomal bupivacaine are injected into the liposomal bupivacaine group
- Standard Bupivacaine: SB (Standard Bupivacaine) group - This group will be receiving 60 mL of 0.25% bupivacaine in total, 30 mL on each side.
  For the QL block, Shamrock sign consistent of the quadratus lumborum muscle, psoas major muscle, erector spinae muscles and the L4 transverse process will be identified. Under ultrasound guidance with an in-plane technique, the needle will be advanced into the fascial plane between the quadratus lumborum and psoas major muscles. Local anesthetic will be injected into the plane.
  Bupivacaine Hydrochloride: 40 mL of 0.125% bupivacaine hydrochloride are injected into the liposomal bupivacaine group.
  60mL of 0.25% bupivacaine hydrochloride are injected into the standard bupivacaine group
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [40 to 69] | 62 [54 to 69] | 61.5 [48 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 24 | 42
  Male | 20 | 16 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 36 | 36 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body Mass Index [Median (Inter-Quartile Range); unit: kg/square meter] | 25.8 [23.6 to 30.1] | 28.7 [24.2 to 33.1] | 26.9 [23.7 to 31.5]
No Known Allergies [Count of Participants; unit: Participants] | 17 | 17 | 34
Height [Median (Inter-Quartile Range); unit: cm] | 172.7 [165.1 to 180.3] | 167.3 [161.0 to 177.8] | 170.2 [162.0 to 178.0]
Weight [Median (Inter-Quartile Range); unit: kg] | 76.8 [68.7 to 93.4] | 77.5 [67.7 to 96.1] | 77.1 [68.4 to 94.4]

OUTCOME MEASURES:

1. Primary Outcome: VAS Score at 1 Hour at Rest
Description: The VAS score at rest will be measured by a study team investigator using Visual Analog Scale (VAS). Using a scale of 1-10 for documentation with 10 being the worst pain and 0 being no pain
Time Frame: Pain scores will be measured 1 hour after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
score on a scale | 5.0 [0.0 to 7.0] | 3.0 [0.0 to 6.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model least squares (LS) means differences with Sidak adjustment for multiple comparisons; p = 0.54, Mixed Models Analysis; Sidak adjustment

2. Primary Outcome: VAS Score at 1 Hour With Movement
Description: The VAS score with movement (knee flexion) will be measured by a study team investigator using Visual Analog Scale (VAS). Using a scale of 1-10 for documentation with 10 being the worst pain and 0 being no pain
Time Frame: Pain scores will be measured 1 hour after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
score on a scale | 5.0 [0.0 to 8.0] | 3.0 [0.0 to 6.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.59, Mixed Models Analysis

3. Primary Outcome: VAS Score at 24 Hours at Rest
Description: as for outcome 1
Time Frame: Pain scores will be measured 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
score on a scale | 4.0 [2.0 to 6.0] | 3.0 [2.0 to 5.5]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.98, Mixed Models Analysis — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; Sidak adjustment

4. Primary Outcome: VAS Score at 24 Hours With Movement
Description: as for outcome 2
Time Frame: Pain scores will be measured 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
score on a scale | 7.0 [4.0 to 9.0] | 6.0 [3.0 to 8.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.94, Mixed Models Analysis — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; Sidak adjustment

5. Primary Outcome: VAS Score at 48 Hours at Rest
Description: as for outcome 1
Time Frame: Pain scores will be measured 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
score on a scale | 3.0 [1.0 to 6.0] | 2.5 [1.0 to 5.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.86, Mixed Models Analysis; Sidak adjustment

6. Primary Outcome: VAS Score at 48 Hours With Movement
Description: as for outcome 2
Time Frame: Pain scores will be measured 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
score on a scale | 5.0 [3.0 to 7.0] | 5.0 [3.0 to 6.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 1.0, Mixed Models Analysis — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; Sidak adjustment

7. Primary Outcome: VAS Score at 72 Hours at Rest
Description: as for outcome 1
Time Frame: Pain scores will be measured 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
score on a scale | 2.0 [0.0 to 4.0] | 2.0 [0.5 to 4.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.99, Mixed Models Analysis

8. Primary Outcome: VAS Score at 72 Hours With Movement
Description: as for outcome 2
Time Frame: Pain scores will be measured 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
score on a scale | 4.0 [2.0 to 6.0] | 3.0 [2.0 to 5.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.99, Mixed Models Analysis

9. Secondary Outcome: Total Opioid Consumption at 1 Hour
Description: Opioid consumption will be collected by a study team member post operatively for 3 days per protocol time requirements
Time Frame: Opioid consumption will be measured at 1 hour post op. The total amount will be recorded
Measure: Median (Inter-Quartile Range); unit: morphine equivalent units
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
morphine equivalent units | 8.0 [0 to 16.0] | 2.0 [0.0 to 15.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.72, Mixed Models Analysis

10. Secondary Outcome: Total Opioid Consumption at 24 Hour
Description: Opioid consumption will be collected by a study team member post operatively for 3 days per protocol time requirements
Time Frame: Opioid consumption will be measured at 24 hour post op. The total amount will be recorded
Measure: Median (Inter-Quartile Range); unit: morphine equivalent units
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
morphine equivalent units | 54.0 [23.0 to 98.5] | 30.0 [5.0 to 62.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.29, Mixed Models Analysis

11. Secondary Outcome: Total Opioid Consumption at 48 Hour
Description: Opioid consumption will be collected by a study team member post operatively for 3 days per protocol time requirements
Time Frame: Opioid consumption will be measured at 48 hour post op. The total amount will be recorded
Measure: Median (Inter-Quartile Range); unit: morphine equivalent units
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
morphine equivalent units | 43.8 [7.5 to 90.0] | 15.0 [5.5 to 45.0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.46, Mixed Models Analysis

12. Secondary Outcome: Total Opioid Consumption at 72 Hour
Description: Opioid consumption will be collected by a study team member post operatively for 3 days per protocol time requirements
Time Frame: Opioid consumption will be measured at 72 hour post op. The total amount will be recorded
Measure: Median (Inter-Quartile Range); unit: morphine equivalent units
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
morphine equivalent units | 17.5 [0.0 to 60.0] | 15.0 [0.0 to 38.8]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard Bupivacaine; Test type: Other — P values are from mixed model LS means differences with Sidak adjustment for multiple comparisons; p = 0.77, Mixed Models Analysis

13. Other Pre Specified Outcome: Nausea Scores (None) at 1 Hour
Description: Nausea scores will be collected by a study team member post operatively up to 3 days per protocol. Nausea will be recorded as none, mild, moderate, or severe
Time Frame: Nausea scores will be measured at 1 hour post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 34 | 38

14. Other Pre Specified Outcome: Nausea Scores (Mild) at 1 Hour
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 1 hour post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 4 | 1

15. Other Pre Specified Outcome: Nausea Scores (Moderate) at 1 Hour
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 1 hour post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 0 | 1

16. Other Pre Specified Outcome: Nausea Scores (Severe) at 1 Hour
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 1 hour post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 0 | 0

17. Other Pre Specified Outcome: Nausea Scores (None) at 24 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 24 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 26 | 27

18. Other Pre Specified Outcome: Nausea Scores (Mild) at 24 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 24 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 5 | 9

19. Other Pre Specified Outcome: Nausea Scores (Moderate) at 24 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 24 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 2 | 3

20. Other Pre Specified Outcome: Nausea Scores (Severe) at 24 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 24 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 2 | 0

21. Other Pre Specified Outcome: Nausea Scores (None) at 48 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 48 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 25 | 28

22. Other Pre Specified Outcome: Nausea Scores (Mild) at 48 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 48 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 5 | 9

23. Other Pre Specified Outcome: Nausea Scores (Moderate) at 48 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 48 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 2 | 3

24. Other Pre Specified Outcome: Nausea Scores (Severe) at 48 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 48 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 6 | 0

25. Other Pre Specified Outcome: Nausea Scores (None) at 72 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 72 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 26 | 29

26. Other Pre Specified Outcome: Nausea Scores (Mild) at 72 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 72 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 7 | 8

27. Other Pre Specified Outcome: Nausea Scores (Moderate) at 72 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 72 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 4 | 3

28. Other Pre Specified Outcome: Nausea Scores (Severe) at 72 Hours
Description: as for outcome 13
Time Frame: Nausea scores will be measured at 72 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 1 | 0

29. Other Pre Specified Outcome: Sedation Scores (Awake/Alert) at 1 Hour
Description: Sedation scores will be collected by a study team member post operatively up to 3 days per protocol requirements. Determining if patient is awake, alert, quietly awake, asleep and arousable, or deep sleep.
Time Frame: Sedation scores will be documented at 1 hour post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 6 | 8

30. Other Pre Specified Outcome: Sedation Scores (Quietly Awake) at 1 Hour
Description: as for outcome 29
Time Frame: Sedation scores will be documented at 1 hour post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 26 | 15

31. Other Pre Specified Outcome: Sedation Scores (Asleep/Arousable) at 1 Hour
Description: as for outcome 29
Time Frame: Sedation scores will be documented at 1 hour post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 19 | 22

32. Other Pre Specified Outcome: Sedation Scores (Deep Sleep) at 1 Hour
Description: as for outcome 29
Time Frame: Sedation scores will be documented at 1 hour post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 3 | 4

33. Other Pre Specified Outcome: Sedation Scores (Awake/Alert) at 24 Hours
Description: as for outcome 29
Time Frame: Sedation scores will be documented at 24 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 36 | 36

34. Other Pre Specified Outcome: Sedation Scores (Awake/Alert) at 48 Hours
Description: as for outcome 29
Time Frame: Sedation scores will be documented at 48 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 35 | 38

35. Other Pre Specified Outcome: Sedation Scores (Awake/Alert) at 72 Hours
Description: as for outcome 29
Time Frame: Sedation scores will be documented at 72 hours post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 36 | 37

36. Other Pre Specified Outcome: Surgery Duration
Description: Duration of surgery will be collected per MR of surgeon documentation.
Time Frame: Duration of Surgery from surgery start time to surgery stop time (usually within 6 hours)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
minutes | 222.5 [157.0 to 285.0] | 222.5 [154.0 to 266.5]

37. Other Pre Specified Outcome: Length of Stay
Description: Admission date until Admission Discharge
Time Frame: Time Frame for Admission to Discharge (usually within 3-7 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
days | 3.5 [2.9 to 4.3] | 3.1 [2.3 to 5.0]

38. Other Pre Specified Outcome: Time to Flatus
Description: Hours for End of Surgery to first reported hour of Flatus
Time Frame: End of Surgery until first reported Flatus (usually within 3 to 5 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
hours | 20.1 [14.3 to 34.7] | 21.5 [15.9 to 37.2]

39. Other Pre Specified Outcome: Time to Bowel Movement
Description: Hours for End of Surgery to first reported hour of bowel movement
Time Frame: End of Surgery until first reported Bowel movement per MR or patient reported (usually 3 to 5 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
hours | 33.0 [17.5 to 61.5] | 26.4 [18.5 to 53.2]

40. Other Pre Specified Outcome: Time to Per Os
Description: Reported time after surgery to time of Os per MR or patient
Time Frame: Time from end of surgery to time of Os (usually 4-16 hours)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
hours | 7.1 [4.4 to 14.2] | 6.6 [3.6 to 11.1]

41. Other Pre Specified Outcome: Ambulatory Postoperatively
Description: Number of patients who ambulated within 24 hours of end of surgery
Time Frame: End of Surgery until first reported ambulated postoperatively per MR or patient reported (Usually within 24 hours postop)
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
Number analyzed (Participants) | 38 | 40
Participants | 35 | 40

ADVERSE EVENTS:
Time Frame: 72 hours postoperative
Arm/Group | Liposomal Bupivacaine | Standard Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT03702621/Prot_SAP_000.pdf